CLINICAL TRIAL: NCT06048497
Title: The Role of Carotid Flow Time-Based Fluid Administration in the Incidence of Hypotension After Spinal Anesthesia in Patients Undergoing Caesarean Section
Brief Title: The Role of Carotid Flow Time-Based Fluid Administration in Caesarean Section
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Demet Laflı Tunay, Principal Investigator, Cukurova University
Other Study IDs: FTCCS
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Spinal Anesthesia; Cesarean Section
Keywords: Cesarean section; Carotid flow time; Preload fluid; Hypotension; Spinal anesthesia
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preload: Patients with baseline FTc < 327 ms were assigned to the preload group, and Ringer Lactate (RL) preload fluid administration to these patients was continued until FTc > 327 ms.
  Interventions: Device: Corrected carotid flow time measurement guided fluid preload
- Non-preload: Patients with baseline FTc > 327 ms were assigned to the non-preload group, and preload fluid was not administered to these patients

INTERVENTIONS:
Device: Corrected carotid flow time measurement guided fluid preload — Preoperative FTcs of pregnant women who underwent C/S operation were measured, and those below the cut-off value (327 ms) determined in previous studies were preloaded with Ringer Lactate until FTc was > 327 ms.
  Groups: Preload

SUMMARY:
It has been reported that corrected carotid flow time (FTc) may indicate the responsiveness of spontaneously breathing patients to fluid therapy. The primary objective of the study is to determine the effect of fluid preload applied to patients with preanesthetic FTc values below the cut-off value on the incidence of hypotension in cesarean section (C/S) surgery. Pregnant women who underwent cesarean section under spinal anesthesia were included in this prospective study. In the preoperative care unit, patients were assigned to two groups according to their baseline FTc values. Patients with baseline FTc < 327 ms were assigned to the first group, and Ringer Lactate (RL) preload fluid administration to these patients was continued until FTc > 327 ms. On the other hand, patients with baseline FTc > 327 ms were assigned to the second group, and preload fluid was not administered to these patients. Intraoperative hemodynamic data were recorded for each patient.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years of age pregnant women
* American Society of Anesthesiologists (ASA) physical status-II patients
* Uncomplicated, singleton, term pregnancy
* Elective C/S surgery

Exclusion Criteria:

* Placental disorders
* Gestational hypertensive disorders
* Morbid obesity (BMI>39 kg/m2)
* Carotid stenosis more than 50%
* Baseline SAP more than 160 mmHg
* Arrhythmia
* History of cardiovascular or cerebrovascular disease, and chronic kidney disease (estimated glomerular filtration rate <60 mL/min/1.73 m2)
* Emergency surgery

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: ASA II pregnant women between the ages of 20 and 40 who were undergoing elective cesarean section, and had uncomplicated singleton term pregnancies, and agreed to participate in the study were included.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
The incidence of intra-operative hypotension | During surgery
  Hypotension definitions included systolic arterial pressure (SAP) below 80 mmHg, or mean arterial pressure (MAP) below 65 mmHg, or a decrease in SAP of more than 30% below baseline, or a decrease in MAP of more than 20% below baseline, or any combination of all these definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Demet Laflı Tunay, Dr., Principal Investigator — Çukurova University, Balcalı Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Cukurova University, Adana, Saricam
  - Çukurova University; Faculty of Medicine, Adana, Sarıçam

IPD SHARING:
Plan to Share IPD: No
All data were anonymized by the local researcher. Therefore, data collection was pseudonymous and the patient's name did not appear on any case report form or other study document. All collected data were kept confidential. This study was conducted in accordance with the revision of the Declaration of Helsinki (2008). International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) was strictly adhered to.